CLINICAL TRIAL: NCT00063258
Title: Phase II Randomized Open-Label Trial of the EGFR Tyrosine Kinase Inhibitor OSI-774 (Tarceva™) in Combination With Paclitaxel and Carboplatin Prior to Surgery in Resectable Stage IIIA (N2) and IIIB (T4 N2) NSCLC: A Clinical Outcome and Biological Endpoint Trial
Brief Title: Tarceva Surgery for Resectable Stage IIIA(N2) and IIIB (T4 N2) Non-Small-Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID02-327
Record Dates: First submitted 2003-06-24; First posted 2003-06-25 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; OSI-774; Tarceva; Carboplatin; Paclitaxel; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + Tarceva (Active Comparator)
  Interventions: Drug: Tarceva (OSI-774); Drug: Paclitaxel; Drug: Carboplatin
- Chemotherapy Alone (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Tarceva (OSI-774) — 150 mg/day, starting day 1 and stopping night prior to surgery.
  Other Names: Tarceva
  Arms: Chemotherapy + Tarceva
Drug: Paclitaxel — Planned dose of 200 mg/m^2 continuous IV infusion over 3 hours on Day 1 of each 21-day cycle.
  Other Names: Taxol
Drug: Carboplatin — Dose of AUC = 6 mg/ml × min began within 60 minutes following completion of paclitaxel infusion, infused over 15-30 minutes on Day 1 of Cycle 1 of each 21-day cycle, and then on Day 1 of each subsequent cycle according to institutional standards.

SUMMARY:
The goal of this clinical research study is to learn about the safety and effectiveness of OSI-774 when combined with standard chemotherapy (carboplatin and paclitaxel) before surgery in the treatment of non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a phase II, single institution open label randomized trial of induction carboplatin and paclitaxel plus/minus daily oral OSI-774 in patients with potentially resectable NSCLC that is stage IIIA and IIIB (T4 satellite nodules or invasion into T4 structures but no malignant effusion.) N3 disease is excluded. Patients will be required to have pathologically demonstrated N2 disease via mediastinoscopy. Forty patients will be treated with 3 courses of chemotherapy followed by surgery. Ten of these patients will be randomized to chemotherapy alone and 30 patients to chemotherapy plus OSI-774. The 10 patients will serve as a chemotherapy alone control for molecular endpoint analysis. OSI-774 will be stopped the night before surgery. At the time of surgery, pathologic response will be determined. Following surgery, patients will be treated with consolidation radiation therapy if there are positive margins or N2 lymph nodes at the time of resection. Patients who have no N2 disease at surgery will have the option of consolidation radiation therapy but will not be required to have it done. Patients not able to tolerate radiation even if they have N2 disease or positive margins at surgery may continue on this study. This will be followed by maintenance OSI-774 for patients from both arms of the study. OSI-774 will be continued as maintenance to a maximum of 2 years following surgery. Tissue for molecular studies will be obtained pretreatment either at the time of diagnostic biopsy or mediastinoscopy. Post-treatment tissue will be obtained at the time of surgery. This tissue will be assayed for defined molecular endpoints using immunohistochemistry, immunoprecipitation and mRNA expression analysis. Blood, urine, hair follicles, and skin samples will also be collected from patients who consent to provide these.

ELIGIBILITY:
Inclusion Criteria:

1. Must have signed consent for LAB03-0383
2. Pathologic documentation of NSCLC
3. Stage IIIA and IIIB (T4 satellite nodules or invasion into T4 structures but no malignant effusion) with all patients requiring mediastinoscopy positive N2, potentially resectable disease. N3 disease is excluded.
4. Measurable disease
5. Zubrod performance status of 0 or 1
6. Calculated post-resectional FEV1 of > 40%
7. WBC>4000/l, ANC>1500/l, platelets > 100,000/l
8. Serum creatinine < 1.5 ULN or calculated creatinine > 50 cc/min
9. Total serum bilirubin <1.5 x ULN or SGPT or SGOT < 2 X ULN
10. The following must be completed within 28 days of registration: CT scan of the chest and upper abdomen to include the adrenals. Mediastinoscopy to document ipsilateral nodal involvement and exclude N3 disease Blood tests, and pulmonary function tests The following must be completed within 2 months of registration: Pet scan If a CT PET is done more than 28 days, only the CT needs to be repeated and a bone scan to rule out bone metastases

Exclusion Criteria:

1. No prior chemotherapy or radiation for NSCLC
2. No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease-free for at least five years. If patient is suspected or known to have basal or squamous skin cancer, this maybe treated after induction chemotherapy is completed at the time of thoracotomy.
3. No post-obstructive pneumonia or other serious infection or other serious underlying medical condition that would impair ability of patient to receive protocol treatment, including prior allergic reactions to drugs containing cremophor.
4. Pregnant or nursing women may not participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Zinner, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 10/13/2003 to 03/18/2008; All patients recruited at University of Texas M.D. Anderson Cancer Center
Pre-assignment Details: Study terminated due to low accrual; No evaluable patients were assigned to Chemotherapy Alone group (anticipated randomization to have been 10 of 40 patients treated with 3 courses of chemotherapy).
Period: Overall Study
Arm/Group | Chemotherapy + Tarceva | Chemotherapy Alone
Started | 5 | 0
Completed | 1 | 0
Not Completed | 4 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy + Tarceva | Chemotherapy Alone | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Continuous [Median (Full Range); unit: years] | 64 [56 to 71] |  | 64 [56 to 71]
Gender [Number; unit: participants]
  Female | 1 |  | 1
  Male | 4 |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response
Description: Response defined by tumor assessment using Response Evaluation Criteria In Solid Tumors (RECIST) to learn effectiveness of Tarceva (OSI-774) when combined with standard chemotherapy before surgery.
Time Frame: 5 Years to collect outcome information
Population: Analysis limited since of 5 participants enrolled, only 1 evaluable for response.
Measure: Number; unit: Participants
Arm/Group | Chemotherapy + Tarceva | Chemotherapy Alone
Number analyzed (Participants) | 1 | 0
Participants
  Complete Response | 0 |
  Partial Response | 0 |
  Stable Disease | 1 |
  Progressive Disease | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study activation (June 17, 2003) to 30 days following last dose of study treatment (approximately 2 years and 5 months)
Arm/Group | Chemotherapy + Tarceva | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 1/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Chemotherapy + Tarceva (N=5) | Chemotherapy Alone (N=0)
Hemoptysis (Grade 1) (Blood and lymphatic system disorders) | 1/1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy + Tarceva (N=5) | Chemotherapy Alone (N=0)
Abdominal Cramping (Grade 2) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alopecia (Grade 2) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bilirubin Increase (Grade 1) (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diarrhea (Grade 3) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Skin (Grade 2) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysphagia (Grade 1) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (Grade 2) (General disorders) | 1 (1) | 0 (0)
Infection Clinical with Grade 3-4 ANC (Wound) (Infections and infestations) | 1 (1) | 0 (0)
Infection with Normal ANC (Bladder -Urinary) Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Infection with Normal ANC (Wound) Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Grade 3) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Grade 1) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Grade 3) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neuropathy: Sensory (Grade 1) (Nervous system disorders) | 1 (1) | 0 (0)
Pain (Grade 2) (General disorders) | 1 (1) | 0 (0)
Palpitations (Grade 3) (Cardiac disorders) | 1 (1) | 0 (0)
Rash/Desquamation (Grade 3) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stomatitis (Grade 2) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Taste Alteration (Grade 2) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Grade 2) (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Despite active study recruitment and screening for this study, only 5 subjects were enrolled out of the planned 40 subjects. Of the 5 subjects enrolled, only 1 patient was evaluable for response assessment. The study was subsequently terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No